CLINICAL TRIAL: NCT05246501
Title: The Effect of The Standardized Patient Simulation Method on Teaching Nursing Students The Skill Of Caring for Individual Diagnosed With Dementia
Brief Title: The Effect of Simulation in Gaining Skills to Nursing Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Aydan Akkurt Yalçıntürk, PHD Student in Nursing Department, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SY200217B06
Record Dates: First submitted 2022-01-11; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Dementia; Nursing Caries
Keywords: Dementia; patient simulation; nursing education; nursing student; simulation training
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation (Experimental)
  Interventions: Other: Simulation
- control group (Active Comparator)
  Interventions: Other: No simulation

INTERVENTIONS:
Other: Simulation — A case scenario with a diagnosis of dementia was used in the study. The scenario consisted of preliminary preparation, implementation and evaluation parts. Psychiatric nursing laboratory practice was applied to the students in the scenario study group. An elderly female standard patient who was diagnosed with dementia took part in the scenario. During this simulation, students were expected to perform mental state examination of the patient, use therapeutic communication techniques and ensure environmental safety.
  Arms: Simulation
Other: No simulation — The students in the control group did not receive simulation training.
  Arms: control group

SUMMARY:
This research is a randomized controlled study conducted to examine the effect of standard patient simulation training in providing nursing students with the ability to care for individuals with dementia.

The population of the research consisted of 100 students who were enrolled in the Nursing Faculty and took the "Psychiatric Nursing" course in 2020-2021 academic year. 84 students who were in the universe and completed the pre-test were randomly assigned to the experimental groups that received simulation training and the control groups that did not receive simulation training. The study was completed with 36 students in the experimental group and 35 students in the control group. Research data were collected with "Personal Coding System and Scale Cover Document", "Structured Student Information Form", "Dementia Information Test", "Case Study Form for Individuals Diagnosed with Dementia", "Standardized Mini Mental Examination", "Communication Skills Evaluation Form", Nursing Diagnosis Detection Skill Form" and "Modified-Simulation Effectiveness Tool".

ELIGIBILITY:
Inclusion Criteria:

* Registered in Hamidiye Faculty of Nursing,
* Taking a psychiatric nursing course in the spring semester of the 2020-2021 academic year,
* Do not have a communication problem at a level that prevents meeting,
* Students who volunteered to participate in the study were included in the study.

Exclusion Criteria:

* Not registered in Hamidiye Nursing Faculty,
* Those who did not take a psychiatric nursing course in the spring semester of the 2020-2021 academic year,
* Having a communication problem at a level that prevents meeting,
* Students who did not volunteer to participate in the study were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Scale Cover Document with Personal Coding System | for three months
  Scale Cover Document with Personal Coding System: A rare code was found with the coding of the first letter of the students' mothers' maiden name, the month of birth, the total number of siblings, the number of sisters, the number of brothers
students' introductory characteristics | before simulation.
  Students were asked to fill in the pretest and posttest.
  Structured Student Information Form: In this form, which was created by scanning the literature, the age, gender, high school graduated, economic status, the presence of a person diagnosed with dementia in the family, the closeness of the individual diagnosed with dementia, the status and duration of living with the individual with dementia, the status and duration of caring for the individual with dementia. There are 12 questions in total, consisting of self-confidence in caregiving, feeling competent and willing, getting information about dementia, sources of information and the first word that comes to mind when dementia is mentioned (Webster and DiBartolo, 2014; Maharaj, 2017).
Dementia Knowledge | for three months
  Dementia Knowledge Test: The Dementia Knowledge Test consists of thirty items prepared by the researchers based on the literature in order to determine the knowledge levels of students on the symptoms, etiology, treatment and nursing care for dementia. (Toye et al., 2014; NICE, 2021; Shaji et al., 2018; Akgün Çıtak, 2016). Students were asked to mark one of the correct, I don't know, incorrect answers for each item. In order to evaluate the test in terms of language, expression, intelligibility, coverage of the subject and whether it contains scientific errors, the opinions of six experts, independent of each other, were taken. The form was rearranged in line with expert opinions.
assessment standardized mini mental test | for three months
  Case Study Form for Individuals Diagnosed with Dementia: The form developed by the researchers consists of four parts for the case study of an individual diagnosed with dementia. In the first part, students were asked to indicate the "Standardized Mini Mental State Test" score for the individual in the case study. In the second part, students were asked to mark one of the statements "I agree", "I am undecided" and "I disagree" for the nursing diagnoses given in accordance with the case. In the third part, they were asked to mark one of the statements "I agree", "I am undecided" or "I disagree" for the nursing interventions specified for the nursing diagnoses of "Lack of self-care", "Risk of trauma" and "Chronic Confusion". In the last section, they were asked to mark one of the statements "I agree", "I am undecided" or "I do not agree" for the items that should be considered when communicating with a person with dementia.
determining a nursing diagnosis | for three months
  Case Study Form for Individuals Diagnosed with Dementia: The form developed by the researchers consists of four parts for the case study of an individual diagnosed with dementia. In the first part, students were asked to indicate the "Standardized Mini Mental State Test" score for the individual in the case study. In the second part, students were asked to mark one of the statements "I agree", "I am undecided" and "I disagree" for the nursing diagnoses given in accordance with the case. In the third part, they were asked to mark one of the statements "I agree", "I am undecided" or "I disagree" for the nursing interventions specified for the nursing diagnoses of "Lack of self-care", "Risk of trauma" and "Chronic Confusion". In the last section, they were asked to mark one of the statements "I agree", "I am undecided" or "I do not agree" for the items that should be considered when communicating with a person with dementia.
identifying nursing interventions | for three months
  Case Study Form for Individuals Diagnosed with Dementia: The form developed by the researchers consists of four parts for the case study of an individual diagnosed with dementia. In the first part, students were asked to indicate the "Standardized Mini Mental State Test" score for the individual in the case study. In the second part, students were asked to mark one of the statements "I agree", "I am undecided" and "I disagree" for the nursing diagnoses given in accordance with the case. In the third part, they were asked to mark one of the statements "I agree", "I am undecided" or "I disagree" for the nursing interventions specified for the nursing diagnoses of "Lack of self-care", "Risk of trauma" and "Chronic Confusion". In the last section, they were asked to mark one of the statements "I agree", "I am undecided" or "I do not agree" for the items that should be considered when communicating with a person with dementia.
be able to apply standardized mini mental test | during simulation.
  standardized mini mental test: Developed by Folstein et al. (1975), the test provides the grading of cognitive disorders and evaluates cognitive functions in five different parts (orientation, registration, attention and calculation, recall, and language) (Folstein et al., 1975). Turkish validity and reliability were determined by Güngen et al. (2002) by The highest score from the test is 30. Orientation questions are 10 points, recording memory and recall 6 points, attention and calculation 5 points, naming 2 points, repetition 1 point, commands 3 points, reading 1 point, writing 1 point, structuring skill 1 point. A score of less than 24 on the Standardized Mini Mental Test (SMMT) indicates dementia, a score of 24-26 indicates mild neurocognitive impairment, and a score of 26 and above indicates normal cognitive functions. SMMT was found to be a valid and reliable tool in patients with mild dementia in our society.
Communication Skills | during simulation.
  Communication Skills Evaluation Form: It was prepared by researchers in line with the literature on the subject (Jootun & McGhee, 2011; Akgün Çıtak, 2016; Dikeç & Kutlu, 2020) in order to objectively evaluate the performance of students regarding communication skills. The form consists of 26 items. The performance of the students, when each step of the student is applied; Evaluated by marking "fully done", "partly done", "did not do"
Things to consider when contacting | for three months
  Case Study Form for Individuals Diagnosed with Dementia: The form developed by the researchers consists of four parts for the case study of an individual diagnosed with dementia. In the first part, students were asked to indicate the "Standardized Mini Mental State Test" score for the individual in the case study. In the second part, students were asked to mark one of the statements "I agree", "I am undecided" and "I disagree" for the nursing diagnoses given in accordance with the case. In the third part, they were asked to mark one of the statements "I agree", "I am undecided" or "I disagree" for the nursing interventions specified for the nursing diagnoses of "Lack of self-care", "Risk of trauma" and "Chronic Confusion". In the last section, they were asked to mark one of the statements "I agree", "I am undecided" or "I do not agree" for the items that should be considered when communicating with a person with dementia (Dilek et al., 2017; Akgün Çıtak, 2016).
Nursing Diagnosis Detection Skill | during simulation.
  Nursing Diagnosis Detection Skill Form: It was prepared with the aim of evaluating students' performance in nursing diagnosis detection skills. Students were asked to write down their nursing diagnoses in accordance with the simulation scenario.
Students' perceptions of the effectiveness of learning in a simulation environment | during simulation
  Modified-Simulation Efficiency Tool: The measurement tool for students' perceptions of the effectiveness of learning in a simulation environment consists of four sub-dimensions, namely preliminary information, learning, trust and analysis, and nineteen items. The Cronbach Alpha internal consistency coefficient of the measurement tool is 0.92. The items of the scale are scored from 1 to 5 as "Strongly Disagree", "Partly Disagree", "Undecided", "Partly Agree" and "Strongly Agree". "Pre-informing" sub-dimension score range is 2-10, "Learning sub-dimension" score range is 4-25, "Confidence" sub-dimension score range is 7-35, and "Analysis" sub-dimension score range is 5-25. The total score is obtained by summing the scores of all sub-dimensions. The score range is between 18 and 95, and a high score indicates that the student's perception of the effectiveness of learning in the simulation environment is positive.

CONTACTS AND LOCATIONS:
Overall Officials: Aydan Akkurt Yalçıntürk, Lecturer, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No